CLINICAL TRIAL: NCT03760926
Title: ULTRA Study: a Feasibility, Prospective, Multicenter, Single-arm Trial of the May Health Device in Transvaginal Ablation of Ovarian Tissue Under ULTRAsound Visualisation in Women With Polycystic Ovary Syndrome (PCOS)
Brief Title: A Trial of the May Health Device in Transvaginal Ablation of Ovarian Tissue Under ULTRAsound Visualization in Women With PCOS Infertility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: May Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: ULTRA
Record Dates: First submitted 2018-11-21; First posted 2018-12-03 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Anovulatory infertility
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- May Health Procedure (Experimental): May Health Procedure performed with use of the May Health Kit intended for transvaginal ablation of ovarian tissue under ultrasound visualization in women with infertility due to polycystic ovary syndrome.
  Interventions: Device: May Health Kit

INTERVENTIONS:
Device: May Health Kit — The intervention consists in the realisation of the May Health Procedure using the May Health Kit, which comprises two elements: a disposable device (May Health Device) and a radiofrequency (RF) energy generator (May Health System). The May Health Device is a short-term invasive device delivered and positioned through the vagina to deliver RF energy inside the ovary in order to ablate ovarian tissue.

SUMMARY:
The objective of this study is to provide preliminary evidence for the safety and effectiveness of the May Health Kit in transvaginal ablation of ovarian tissue under ultrasound visualization in women with infertility due to polycystic ovary syndrome.

ELIGIBILITY:
Candidates for this study must meet ALL of the following criteria:

Inclusion criteria for female participants:

1. Age: ≥ 18 to ≤ 40 years
2. Diagnostic of PCOS confirmed by at least 2 of 3 Rotterdam criteria, defined as:

   2.1 Infertility associated with chronic anovulation or oligomenorrhea, defined as spontaneous intermenstrual periods of ≥35 days or a total of ≤9 menses per year 2.2 Ultrasonographic evidence of PCOS (ovarian volume ≥ 10ml and/or follicle number per ovary of ≥ 20) 2.3 Evidence of hyperandrogenaemia: either clinical (hirsutism or acne) or biochemical (raised serum concentration of androgens (testosterone ≥ 2.5nmol/l, or FAI > 4)
3. Ovarian accessibility: determined by ability to bring transvaginal ultrasound transducer into close proximity to ovaries
4. Resistance to first-line pharmacological treatment, defined as at least 2 consecutive non-ovulatory cycles, including at least 1 cycle at the highest dose deemed clinically relevant for the patient
5. At least one patent tube and normal uterine cavity as determined by sonohysterogram, hysterosalpingogram, or hysteroscopy/laparoscopy within the last 3 years
6. Willing to comply with protocol-specified follow-up evaluation
7. Signed informed consent

   Couple inclusion criteria:
8. Normal sperm parameters based on WHO 2000 criteria (concentration⩾ 15 million/mL, motility A+B ⩾ 32%, normal forms ⩾ 4%).
9. Ability to have regular intercourse during the study
10. No previous sterilization procedures (vasectomy, tubal ligation) that have been reversed

Candidates will be excluded from the study if ANY of the following conditions apply:

1. Pregnant, parturient or breastfeeding women
2. Marked obesity, BMI > 35
3. Marked hyperandrogenism (FAI > 15)
4. Previous ovarian surgery: LOD, endometriosis surgery, ovarian cysts surgery, patients with known or suspected periovarian adhesions.
5. Subject with pacemaker, defibrillator or other active implant
6. Subject is currently participating in another investigational drug or device study that clinically interferes with the endpoints of this study
7. Lack of capacity to give informed consent (individuals deprived of their liberty subject to a legal protection measure or who are unable to express their consent, individuals under guardianship or curatorship)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2023-09-02 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) in terms of type (device/procedure related), seriousness, level of severity. Rate of occurence of intra-procedural and post-procedural adverse events, and device related complications | Up to 30 days
Successful completion of a complete ovarian tissue ablation procedure, which is defined as achievement of the desired number of ablations within each ovary under ultrasound visualization. | During procedure

SECONDARY OUTCOMES:
Occurrence of ovulation following the procedure | Up to 3 months after procedure

OTHER OUTCOMES:
Pain level using the Visual Analogue Scale (VAS - 0 : no pain - 10 : worse pain possible), record of pain medications with doses administered during procedure | At procedure, 7 days, 30 days
Usability of the May Health Kit | During procedure
Pain level using the Visual Analogue Scale (VAS - 0 : no pain - 10 : worse pain possible), record of pain medications with doses administered post-procedure | At 30 days
May Health Procedure time | During procedure
Occurrence of ovulation following the procedure | Up to 6 months after procedure
Pregnancy | At 3, 6, 9 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Saad Amer, MD, PhD, Study Director — Derby Royal Hospital
Locations (6):
- Belgium (2):
  - CHU Saint-Pierre, Brussels
  - CU Saint-Luc, Brussels
- Bicetre Hospital, Le Kremlin-Bicêtre, France
- United Kingdom (3):
  - Royal Derby Hospital, Derby
  - Liverpool Women Hospital, Liverpool
  - Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: No